CLINICAL TRIAL: NCT07146217
Title: An Open-Label, Single-Arm, Pharmacokinetic and Safety Study of Likmez® (Metronidazole Oral Suspension) in Pediatric Patients Aged 12 Months to <4 Years With Anaerobic Bacterial Infection
Brief Title: Pharmacokinetic and Safety Study of Metronidazole Oral Suspension in Pediatric Patients With Anaerobic Bacterial Infection
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Saptalis Pharmaceuticals LLC (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-1501-0X
Record Dates: First submitted 2025-08-08; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Bacterial Infections
Keywords: Anaerobic Bacterial Infection
MeSH Terms: conditions — Bacterial Infections | interventions — Metronidazole; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Likmez® (metronidazole) Oral Suspension (Experimental)
  Interventions: Drug: Likmez® (metronidazole) Oral Suspension

INTERVENTIONS:
Drug: Likmez® (metronidazole) Oral Suspension — Each patient will receive 7.5 mg/kg of Likmez® every 6 hours, with a concentration of 100 mg metronidazole/mL

SUMMARY:
This is an open-label, single-arm, pharmacokinetic and safety study of Likmez® in pediatric patients aged 12 months to <4 years with anaerobic bacterial infection

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 12 months and < 4 years till the time of dosing in the study
* Sufficient venous access to permit cannulation for required blood sample collection.
* Ability to swallow oral liquids.
* Clinical diagnosis with suspected or culture-confirmed anaerobic bacterial infection with pathogens known to be sensitive to metronidazole and requiring treatment for any of the below mentioned infections:

  1. Septicaemia and Bacteraemia
  2. Intra-abdominal infections (including peritonitis, intra-abdominal abscess, and liver abscess)
  3. Bone and joint infections (including osteomyelitis)
  4. Lower respiratory tract infections (including pneumonia, empyema, and lung abscess)
* Patients with clinical diagnosis of polymicrobial infection who can be administered Likmez® with other antibacterial agents without clinically significant drug-drug interactions. Note: These patients will be allowed concomitant administration with other antibacterial drugs, not having an interaction with metronidazole (Refer APPENDIX B: List of Antibiotic Drugs Having Interaction with Metronidazole, for the list of antibiotic drugs having interaction with metronidazole). If co-administration of such medications cannot be avoided, PI should consider taking steps to minimize the risk of QT/QTc interval prolongation and torsade de pointes (TdP), such as electrolyte monitoring and repletion, and ECG monitoring, especially in patients with additional risk factors for TdP.
* Any of the above mentioned clinical conditions, which would allow them to initiate the treatment with IV or oral anti-bacterial drugs with activity against anaerobic bacteria (e.g., IV treatment such as a betalactam/beta-lactamase inhibitor or a cephalosporin plus metronidazole; or oral treatment such as amoxicillin, amoxicillin-clavulanate, or azithromycin) followed by treatment with i.e. Likmez® at 7.5 mg/kg, to complete the treatment course and are able to provide PK samples for the study.
* Parents/legal guardians of the patient have provided Written Informed Consent prior to initiation of any protocol-specific procedures.

Exclusion Criteria:

* History of anaphylactic reaction to metronidazole or other nitroimidazole derivatives (e.g., tinidazole).
* Presence of clinically significant encephalopathy or peripheral neuropathy.
* Presence or history of clinically significant convulsive seizure disorders.
* Presence or history of any hematologic condition or blood dyscrasia which may result in leukopenia (even if leukocyte count is normal at screening).
* Abnormal laboratory results for the following analyses showing any of the following abnormal results:

  1. Aspartate aminotransferase (AST), alanine transaminase (ALT)>2 X the upper limit of the reference range
  2. WBC count <3.0 X 109 /L
  3. Total bilirubin ≥20 μmol/L (1.17 mg/dL); except in patients with isolated elevation of indirect bilirubin relating to Gilbert syndrome
  4. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 using the Bedside Schwartz methods for estimation (eGFR = 41.3 x height/serum creatinine (Scr), where height is in meters and Scr in mg/dL)
  5. Hemoglobin <8 g/dL
  6. Platelets <100,000/μL
* History or presence of any clinically significant disease or disorder that, in the opinion of the investigator, would put the patient at risk or would potentially influence the results of the study (e.g. evidence of gastrointestinal, hepatic, or renal disease that could affect absorption, distribution, metabolism, or excretion of the orally administered study drug).
* Patients with a history of hereditary fructose intolerance (HFI) or rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency.
* Patients with a known sensitivity to glucose (e.g. patients with a diagnosis of diabetes or patients taking a ketogenic diet).
* Patients with a history of Severe cutaneous adverse reactions (SCARs), including Stevens Johnson syndrome (SJS), Toxic epidermal necrolysis (TEN), drug reaction with eosinophilia and systemic symptoms (DRESS), and acute generalized exanthematous pustulosis (AGEP).
* Patients who have used disulfiram within the last two weeks prior to enrollment in study.
* Patients who have consumed products containing propylene glycol within a week prior to enrollment in study and who wish to continue products containing propylene glycol during the study and for at least three days after the end of treatment period.
* Patients with known status of Cockayne syndrome.
* Patients with treatment with any another drug that is known to have pharmacokinetic interaction [For example: barbiturates such as phenytoin or phenobarbital] with metronidazole, within 30 days prior to enrollment or within 5.5 half-lives of the drug, (whichever is longer), until the end of study.
* Previous exposure to metronidazole within 30 days of enrollment.
* Patients with a known history of Hepatitis B virus (HBV), Hepatitis C virus (HCV), Human immunodeficiency virus (HIV), and latent tuberculosis (TB) infections.
* Previous participation in this study.

Ages: 12 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration [Cmax] | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
  Pharmacokinetic profile of metronidazole and hydroxy-metronidazole (primary metabolite) measured by Cmax
Time to reach at maximum plasma concentration [Tmax] | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
  Pharmacokinetic profile of metronidazole and hydroxy-metronidazole (primary metabolite) measured by Tmax
Area under the concentration-time curve from time 0 to time 't' '[AUC0-t] | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
  Pharmacokinetic profile of metronidazole and hydroxy-metronidazole (primary metabolite) measured by AUC0-t
Volume of distribution [Vd/F] | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
  Pharmacokinetic profile of metronidazole and hydroxy-metronidazole (primary metabolite) measured by Vd/F
Apparent clearance of drug from plasma [CLTotal/F] | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
  Pharmacokinetic profile of metronidazole and hydroxy-metronidazole (primary metabolite) measured by CLTotal/F. The CLTotal will be calculated by dividing the dose by the AUC for the given dosing interval [Dose/ AUC0-Tau]

SECONDARY OUTCOMES:
Comparison of AUC0-t in Pediatric Patients Without Prior IV Metronidazole to Adult Single-Dose PK Data | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
Comparison of Cmax in Pediatric Patients Without Prior IV Metronidazole to Adult Single-Dose PK Data | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
Comparison of AUC0-t in Pediatric Patients With Prior IV Metronidazole to Adult Steady-State PK Data | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
Comparison of Cmax in Pediatric Patients With Prior IV Metronidazole to Adult Steady-State PK Data | Day 1 at Pre-dose (0.00 hour, within 01 hour prior to dosing) and at 01.00, 02.00, 4.00 and 6.00 hours post-dose
Number of Participants With Adverse Events as Assessed by CTCAE v5.0 | From screening to end of study, up to 26 days
Number of Participants with Changes in Systolic Blood Pressure and Diastolic Blood Pressure | From screening to end of study, up to 26 days
Number of Participants with Changes in Respiratory Rate | From screening to end of study, up to 26 days
Number of Participants with Changes in Pulse Rate | From screening to end of study, up to 26 days
Number of Participants with Changes in Body Temperature | From screening to end of study, up to 26 days
Number of Participants with Changes of P wave in Electrocardiogram (ECG) | From screening to end of study, up to 26 days
Number of Participants with Changes of QRS complex in Electrocardiogram (ECG) | From screening to end of study, up to 26 days
Number of Participants with Changes of T wave in Electrocardiogram (ECG) | From screening to end of study, up to 26 days
Number of Participants with Changes in Clinical Laboratory Values | From screening to end of study, up to 26 days
Number of Participants With Abnormal Physical Examination Findings | From screening to end of study, up to 26 days

CONTACTS AND LOCATIONS:
Overall Officials: Polireddy Dondeti, PhD, Study Chair — President & CEO
Locations (3):
- United States (3):
  - Bioresearch Partner, Miami, Florida
  - Empire Medical Clinical Trials, Miami, Florida
  - Aavon Clinical Trials, Richmond, Texas

IPD SHARING:
Plan to Share IPD: Undecided